CLINICAL TRIAL: NCT01758575
Title: Clinical Evaluation of the Underlying Mechanisms of Targeted Therapy Related Toxicities
Status: Terminated | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, H.M.W. Verheul, Prof. dr., Amsterdam UMC, location VUmc
Other Study IDs: 2012/76; 2011-005309-57 (EudraCT Number)
Record Dates: First submitted 2012-12-11; First posted 2013-01-01 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Advanced or Metastatic Solid Malignancy
Keywords: Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and blind biopsies of the oral mucosa, skin and colon mucosa will be taken pre-treatment and after 4 weeks of treatment.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- antiangiogenic tyrosine kinase inhibitors: Sunitinib: 50 mg orally once daily Sorafenib: 400 mg orally twice daily Pazopanib: 800 mg orally once daily
- EGFR inhibitors: Cetuximab 250 mg/m2 intravenously, weekly Panitumumab 6 mg/Kg intravenously, every 2 weeks
- mTOR inhibitors: Everolimus 10 mg orally once daily
- BRAF inhibitor: Vemurafenib 960 mg orally twice daily
- anti-CTL4 antibody: Ipilimumab 3 mg/kg intravenously, every 3 weeks

SUMMARY:
Single center, non-randomized, interventional pilot study with feasibility analysis after enrollment of 20 patients. Adult patients with advanced solid tumors, for whom standard palliative treatment with targeted agents as monotherapy is indicated, including antiangiogenic tyrosine kinase inhibitors, EGFR inhibitors, mTOR inhibitors, BRAF inhibitors and ipilimumab.After feasibility analysis in the first twenty patients, twenty more patients will be included in each of the five drug cohorts. Biopsies will be performed to determine possible immunohistochemical and histopathological changes in normal tissue, possible immunomodulatory changes as expressed by Tcell phenotyping and cytokine profiling and to compare tissue (phospho) proteomic and kinase activity profiles before and during therapy and also at the development of toxicity.The main objective of this pilot study is to determine the biological impact of treatment with targeted agents at the systemic and local tissue level in relation to toxicity.

DETAILED DESCRIPTION:
Rationale: In the past decade multiple agents targeting specific signaling proteins important for tumor growth, including (tyrosine) kinase inhibitors, EGFR inhibitors, mTOR inhibitors and BRAF inhibitors, or agents that modulate the immune response such as ipilimumab, have been developed and have reached clinical approval. Initially it was anticipated that these agents would be active without causing major toxicities, but recent clinical experiences have changed these expectations. Diagnostic tools to predict whether a patient will develop toxicity to targeted agents are not yet available. Our general hypothesis is that immunophenotyping studies combined with (phospho) proteomic and kinase activity profiling in normal tissue before and during treatment with targeted agents may provide more insight in underlying causative mechanisms of toxicity and provide potential biomarkers for clinical use to predict for toxicity.

The investigators hypothesize that targeted therapy- induced toxicity is caused by interference with normal physiological homeostasis at the tissue level. To date, preclinical strategies to predict for clinical toxicities of targeting therapies are lacking.

This study is intended to (1) explore the biological (immunological) mechanisms of targeted agents at the systemic and local tissue level in relation to toxicity (2) determine if off-target receptor kinase inhibition in normal cells and tissues is related to toxicity of the treatment and (3) try to identify novel biomarker(s) predictive of toxicity.

Objective: The main objective of this pilot study is to determine the biological impact of treatment with targeted agents at the systemic and local tissue level in relation to toxicity.

Study design: Single center, non-randomized, interventional pilot study with feasibility analysis after enrollment of 20 patients.

Study population: Adult patients with advanced solid tumors, for whom standard palliative treatment with targeted agents as monotherapy is indicated, including antiangiogenic tyrosine kinase inhibitors, EGFR inhibitors, mTOR inhibitors, BRAF inhibitors and ipilimumab.

Intervention: Patients will be treated with targeted therapies according to the clinical standard guidelines. At this point, five targeted therapies with considerable skin and gastrointestinal toxicities have reached widespread clinical use and therefore "antiangiogenic" tyrosine kinase inhibitors, EGFR inhibitors, mTOR inhibitors, BRAF inhibitors and ipilimumab will be investigated in this study. After feasibility analysis in the first twenty patients, twenty more patients will be included in each of the five drug cohorts. Biopsies will be performed to determine possible immunohistochemical and histopathological changes in normal tissue, possible immunomodulatory changes as expressed by Tcell phenotyping and cytokine profiling and to compare tissue (phospho) proteomic and kinase activity profiles before and during therapy and also at the development of toxicity.

Main study parameters/endpoints: The main objective is to explore the biological impact of treatment with targeted agents at the systemic and local tissue level in relation to toxicity. This objective will be assessed by studying in normal tissue whether treatment with targeted agents induces significant changes in normal tissue of (1) histopathology, such as differences in the presence of infiltrating immune cells, (2) (phospho)proteomic profiles and (3) kinase activity profiles. Secondary objectives are (1) to perform pharmacokinetics and to study whether serum peptide profiles and systemic circulating immune cells and cytokine profiles in patients during treatment with targeted agents are related to toxicity and (2) to identify novel biomarkers predictive of treatment induced toxicity based on pretreatment systemic or local tissue phenotypes.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Enrolment in this study is possible when the indication to receive standard targeted therapy has been determined. Adverse events as a result of this standard treatment may occur. Biopsies of skin, oral mucosa, colon mucosa once prior to and during treatment will be taken. If toxicity develops, a re-biopsy of the affected area will be taken. These biopsies may cause physical discomfort. During therapy, follow-up will include laboratory analysis on a visit to the outpatient clinic. Results of this study may provide new clues for prediction and treatment of targeted therapy induced toxicity

ELIGIBILITY:
Inclusion Criteria:

1. Patients that will start palliative treatment with TKIs, mTOR inhibitors, ipilimumab, vemurafenib or EGFR inhibitors and therefore fulfill according to their attending physician all the usual criteria for receiving standard targeted therapy as monotherapy.
2. PT-INR/PTT < 1.5 x ULN.
3. Platelet count >/= 100 x 109/l

Exclusion Criteria:

1. Concomitant use of anticoagulants
2. Previous colonic surgery in the last 3 months
3. History of inflammatory bowel disease, or other active gastrointestinal infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced or metastatic solid malignancy, amenable to standard treatment with targeted agents will be included from the VUmc Medical Oncology outpatient clinic.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-11; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
histopathological and immunomodulatory changes | 4 weeks
  Biopsies of the areas most anticipated to be affected (skin, oral mucosa, colon mucosa) will be taken at the beginning and after 4 weeks of treatment. Specific attention will be directed in normal tissues at the percentage and types of inflammatory cells and cytokines. In addition, markers of proliferation and apoptosis will be evaluated.
Kinase activity profiles | 4 weeks
  Kinase activity profiles will be measured according to standard methods as developed and modified in the laboratory of VUmc. PamChip will be applied to measure the signal intensity of both the pre- and on- treatment lysates, in the same experiment, to secure comparable conditions. The percentage inhibition is calculated by dividing the mean signal intensity of the on-treatment lysate by the mean signal intensity of the pre-treatment normal tissue lysates.
Kinome wide and quantitative (phospho)proteomic profiles | 4 weeks
  Kinome wide and quantitative (phospho)proteomic profiles will be determined in normal tissue biopsies before and during treatment, for each patient. We anticipate that these profiles will reveal information on the effect of treatment on kinase abundances, phosphopeptide levels and on phosphorylation sites. Differences in levels of phosphopeptides and fold-change of phosphorylation sites will be quantified. We will try to correlate observed profile changes to toxicity development.

SECONDARY OUTCOMES:
Based on the results of the primary aim, potential novel markers predictive for toxicity will be evaluated using the measurements as described under the primary subaims 1-3 | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Henk MW Verheul, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands